CLINICAL TRIAL: NCT05602974
Title: Adjuvant Stereotactic Body Radiotherapy (SBRT) for Hepatocellular Carcinoma After Hepatectomy With Narrow Margin: a Prospective, Multicenter, Randomized Controlled, Open-labelled, Phase III Study
Brief Title: Adjuvant Stereotactic Body Radiotherapy (SBRT) for Hepatocellular Carcinoma After Hepatectomy With Narrow Margin: a Prospective, Multi-center, Randomized Controlled, Open-labelled, Phase III Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0908
Record Dates: First submitted 2022-10-29; First posted 2022-11-02 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma; Narrow Margin; Adjuvant Stereotactic Body Radiotherapy; Hepatectomy
Keywords: Hepatocellular carcinoma; Narrow margin; Adjuvant Stereotactic Body Radiotherapy; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Experimental: adjuvant stereotactic body radiation therapy after hepatectomy with narrow margin Control: regular follow-up after hepatectomy with narrow margin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adjuvant stereotactic body radiation therapy (Experimental): adjuvant stereotactic body radiation therapy after hepatectomy with narrow margin
  Interventions: Radiation: stereotactic body radiation therapy
- regular follow-up (Active Comparator): regular follow-up after hepatectomy with narrow margin
  Interventions: Other: regular follow-up

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — adjuvant stereotactic body radiation therapy
  Arms: adjuvant stereotactic body radiation therapy
Other: regular follow-up — regular follow-up
  Arms: regular follow-up

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth prevalent malignancy worldwide. Although surgical excision is considered the standard treatment for resectable HCC, a high rate of postoperative recurrence was observed after partial hepatectomy, with a marginal recurrence rate up to 30%. Narrow margin resection may be the most appropriate procedure for centrally located HCC or HCC located near liver capsule because the premise for survival is the conservation of more normal liver parenchyma. Unfortunately, narrow margin resection has been reported to contribute to poor survival outcomes. However, no adjuvant therapy after hepatectomy is generally considered to be effective in reducing post-operative recurrence.

Radiotherapy (RT) has been well used in many solid malignant tumors as an (neo)adjuvant to surgical treatment, including HCC. SBRT has shown encouraging rates of local control for HCC. Compared with standard fractionation radiation, SBRT can achieve more precise delivery of high-dose radiation beams to the lesion, obtaining a much smaller target volume. Meanwhile, it could be finished in a short period which can bring more convenience to patients. Recently, several study and randomized controlled trials revealed the survival benefit of adjuvant RT (IMRT and SBRT) in patients with HCC. A large-sample and high-quality multi-center, randomized controlled, prospective study is warranted to further confirm the efficacy of adjuvant radiotherapy in patients with narrow margin resection, considering the small sample size of above-mentioned studies.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth prevalent malignancy worldwide. Although surgical excision is considered the standard treatment for resectable HCC, a high rate of postoperative recurrence was observed after partial hepatectomy, with a marginal recurrence rate up to 30%. Narrow margin resection may be the most appropriate procedure for centrally located HCC or HCC located near liver capsule because the premise for survival is the conservation of more normal liver parenchyma. Unfortunately, narrow margin resection has been reported to contribute to poor survival outcomes. However, no adjuvant therapy after hepatectomy is generally considered to be effective in reducing post-operative recurrence.

Radiotherapy (RT) has been well used in many solid malignant tumors as an (neo)adjuvant to surgical treatment, including HCC. SBRT has shown encouraging rates of local control for HCC. Compared with standard fractionation radiation, SBRT can achieve more precise delivery of high-dose radiation beams to the lesion, obtaining a much smaller target volume. Meanwhile, it could be finished in a short period which can bring more convenience to patients. Recently, several study and randomized controlled trials revealed the survival benefit of adjuvant RT (IMRT and SBRT) in patients with HCC. A large-sample and high-quality multi-center, randomized controlled, prospective study is warranted to further confirm the efficacy of adjuvant radiotherapy in patients with narrow margin resection, considering the small sample size of above-mentioned studies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Confirmed diagnosis of HCC. The diagnosis can be established radiographically by the criteria of the American Association for the Study of the Liver (AASLD), or by histologic diagnosis from the core biopsy;
3. Pathologically confirmed as narrow margin (the shortest distance from the edge of the tumor to the surface of liver transection <1cm) ;
4. Child-Pugh class A and B7;
5. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1;
6. Willing to provide tissue from an excisional biopsy of a tumor lesion;
7. For patients with active HBV: HBV DNA < 2000 IU/mL during screening, and have initiated anti-HBV treatment at least 7 days prior to SBRT and willingness to continue anti-HBV treatment during the study;
8. Adequate organ and marrow function as defined below:

1)Marrow: absolute neutrophil count ≥1.5×109/L; platelets ≥50×109/L; hemoglobin ≥90g/L; 2)Liver: total bilirubin ≤3× institutional upper limit of normal (ULN); AST(aspartate aminotransferase) or ALT(alanine aminotransferase) ≤ 5× institutional ULN; albumin ≥29g/L; 3)Kidney: creatinine ≤ 1.5× institutional ULN or estimated glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 (according to the Cockcroft-Gault formula); 9. Women of childbearing potential must be willing to use a highly effective method of contraception for the course of the study through 30 days after radiotherapy. Female patient of childbearing potential should have a negative serum pregnancy test before 72h of her first treatment. Sexually active males must agree to use an adequate method of contraception starting with the treatment through 4 months after radiotherapy.

Exclusion Criteria:

1. Have received radiotherapy for the area to be treated in the past;
2. Severe bleeding tendency or coagulation dysfunction within the previous 6 months;
3. Extrahepatic metastasis;
4. Known history of active Bacillus Tuberculosis (TB)
5. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
6. Active infection requiring systemic therapy;
7. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy;
8. Known psychiatric or substance abuse disorders ;
9. Pregnant or breastfeeding;
10. Known history of human immunodeficiency virus (HIV: HIV 1/2 antibodies);
11. Received a live vaccine within 30 days before radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
marginal recurrence rate | from date of enrollment to date of first documented marginal recurrence. Assessed up to 12 months
  1-year marginal recurrence rate

SECONDARY OUTCOMES:
Overall survival | from date of enrollment to the date of death from any cause. Assessed up to 36 months
  3-year Overall survival
Recurrence free survival | from date of enrollment to the date of first documented recurrence. Assessed up to 36 months
  3-year Recurrence free survival
Time to Progress | from date of enrollment to the date of progress. Assessed up to 36 months
  from date of enrollment to the date of progress. Assessed up to 36 months
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months after SBRT
  Incidence of Treatment-Emergent Adverse events (CTCAE v5.0)
Quality of life by EORTC QLQ-C30 | through study completion, an average of 3 year
  Quality of life by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, MD/PhD, Principal Investigator — Zhejiang University; Weilin Wang, MD/PhD, Principal Investigator — Zhejiang University
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided